CLINICAL TRIAL: NCT06494059
Title: A Novel Repetitive Synchronized Associative Stimulation Neuromodulation Approach for Spinal Cord Injury Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Matija Milosevic, Assistant Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20240454
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: SCI - Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Upper-limb (arms) target group (Experimental): Quadriplegic individuals with SCI who are primary non-ambulatory (walking) will be in this group for up to 2 months.
  Interventions: Other: Intermittent theta burst stimulation (iTBS); Other: Functional electrical stimulation (FES); Other: Transcutaneous spinal cord stimulation (TSCS); Other: Sham Intermittent theta burst stimulation (iTBS)
- Lower-limb (legs) target group (Experimental): Quadriplegic or paraplegic individuals with SCI primary who can walk will be in this group for up to 2 months.
  Interventions: Other: Intermittent theta burst stimulation (iTBS); Other: Functional electrical stimulation (FES); Other: Transcutaneous spinal cord stimulation (TSCS); Other: Sham Intermittent theta burst stimulation (iTBS)
- Trunk (torso) target group (Experimental): Quadriplegic or paraplegic individuals with SCI who are primary wheelchair users will be in this group for up to 2 months.
  Interventions: Other: Intermittent theta burst stimulation (iTBS); Other: Functional electrical stimulation (FES); Other: Transcutaneous spinal cord stimulation (TSCS); Other: Sham Intermittent theta burst stimulation (iTBS)
- Able-bodied target group (Active Comparator): Individuals with no spinal cord injury will be in this group for up to 2 months.
  Interventions: Other: Intermittent theta burst stimulation (iTBS); Other: Functional electrical stimulation (FES); Other: Transcutaneous spinal cord stimulation (TSCS); Other: Sham Intermittent theta burst stimulation (iTBS)

INTERVENTIONS:
Other: Intermittent theta burst stimulation (iTBS) — iTBS is a magnetic stimulation applied using a magnetic coil that is placed on top of the participants head to activate the brain. It consists of three very rapid bursts of electrical pulses at a frequency of 50 Hz (per burst) delivered at a rate of 5 per second for 2 seconds (10 bursts). The burst of pulses will be repeated every 10 seconds for a total duration of about 3 minutes. The stimulation will be applied to activate the brain regions that control upper limb, lower limb or trunk muscles. Each subject is expected to participate longitudinally at least 9 times over 2 months. Each visit will take approximately 2-3 hours.
Other: Functional electrical stimulation (FES) — FES is applied using electrodes that stick to the skin over the muscles or nerves. It will will be applied using an electrical stimulator to produce movements of the hand, leg or the trunk. The stimulation intensity will be determined by gradually increasing strength from 20-100 hertz (hz) until the right amount of movement is obtained. Each subject is expected to participate longitudinally at least 9 times over 2 months. Each visit will take approximately 2-3 hours.
Other: Transcutaneous spinal cord stimulation (TSCS) — TSCS is applied using electrodes that stick to the skin over the spinal cord to activate spinal cord. Mild electrical stimulation will be applied to make sure the nerves on the back are activated (switched on). Different stimulation intensities (strength) will be tested at different frequencies (pulses per second) to determine the best setting for activating the nerves on the back. The stimulus current strength will be adjusted between 0-250 milliamperes (mA) and will remain within the self-reported tolerance limit of each participant. Each subject is expected to participate longitudinally at least 9 times over 2 months. Each visit will take approximately 2-3 hours.
Other: Sham Intermittent theta burst stimulation (iTBS) — Subjects will be fitted with a magnetic coil that is placed on top of the head that does not deliver any stimulation to the brain. Each subject is expected to participate longitudinally at least 9 times over 2 months.Each visit will take approximately 2-3 hours.

SUMMARY:
The purpose of this research is to explore the effect of magnetic stimulation to activate the brain, electrical spinal cord stimulation to activate spinal cord, and electrical muscle stimulation used to activate upper limb (arms), lower limb (legs) and trunk (stomach) muscles in people with spinal cord injury (SCI) and able-bodied subjects (without SCI).

ELIGIBILITY:
Inclusion Criteria:

Male or Female subjects

1. At least 18 years old and no older than 70 years old at the time of enrollment.
2. Able-bodied subjects
3. Traumatic spinal cord injury
4. Upper limb target: neurological level at or above Thoracic 1 level, Abbreviated Injury Scale (AIS) B, C or D impairment grade, primary non-ambulatory;

   * Lower limb target: neurological level at or above Thoracic 10 level, with residual lower limb function; AIS B, C or D impairment grade primary could ambulate;
   * Trunk target: neurological at or above Thoracic 5, AIS A, B, C or D impairment grade, primary wheelchair user
5. Spinal cord injury sustained more than 6 months prior to study.
6. Movement/excitability/etc:

   * Upper limb target: Has detectable residual connection in upper-limb muscles in at least one side confirmed by voluntary electromyography (EMG) or detectable motor evoked potential (MEP) and a visible contraction when functional electrical stimulation (FES) is applied in the hand or wrist muscle at baseline.
   * Lower limb target: Has detectable residual connection in lower-limb muscles in at least one side confirmed by voluntary EMG or detectable MEP and a visible contraction when FES is applied in lower limb ankle plantar or dorsiflexor muscle at baseline.
   * Trunk target: Has detectable residual connection in trunk muscles in at least one side confirmed by voluntary EMG or detectable MEP and a visible contraction when FES is applied in trunk muscle at baseline.
7. Able to commit to intervention and assessment sessions over a maximum duration of 2 months.

Exclusion Criteria:

1. Has traumatic brain injury, stroke, multiple sclerosis, or other disorders that could affect neuromotor function.
2. Has severe spasticity that could prevent the study protocol as determined by the investigator.
3. Has major executive dysfunction, dementia, depression, neurocognitive impairments, or other major medical co-morbidities.
4. Has contraindications for transcutaneous stimulation using FES or TSCS such as breakdown of skin in the area that will come into contact with electrodes, thrombosis, or skin disease.
5. Has a poorly managed autonomic dysreflexia that could be triggered by transcranial magnetic stimulation (TMS), FES, or TSCS.
6. Has a history of prior intracranial surgery or known medical risks that would limit TMS protocols.
7. Has a history of epilepsy, convulsion or seizures.
8. Individuals with metal implants in their head or spine near the sites to be stimulated and other implantable devices (e.g., cochlear implants) in the body that could be affected by TMS or TSCS.
9. Has implanted neurostimulator (e.g., deep brain stimulation (DBS), epidural/subdural, vagal nerve stimulation or VNS).
10. Has a cardiac pacemaker or intracardiac lines.
11. Has peripheral neuropathy, including diabetic polyneuropathy and entrapment neuropathy.
12. Has urinary tract infection, unhealed fracture, contracture, and pressure sore as determined by Braden Scale value of 14 and below.
13. Individuals who require therapy or other care that could interfere with participation in the study.
14. Individuals on investigational drugs or any other intervention known to have a potential impact on neuromotor function.
15. Individuals with substance disorders, including alcoholism and drug abuse.
16. Individuals who are pregnant, breastfeeding, or the desire to become pregnant during the study.
17. In the opinion of the investigators, the study is not safe or appropriate for the participant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in nine-hole peg test | baseline, up to 2 months
  The Nine-Hole Peg Test assesses hand and finger dexterity. It is administered by asking the subject to take the pegs from a container, one by one, and place them into holes on the board as quickly as possible. Participants must then remove the pegs from the holes, one by one, and replace them back into the container. Scores are based on the time taken to complete the activity, recorded in seconds.
Change in foot tapping test (FTT) | baseline, up to 2 months
  FTT assesses motor neuron function and mobility. Participants are seated with the foot on the floor and are asked to tap their foot on the ground as rapidly as possible for 10 seconds while keeping the heel on the ground. The number of taps are counted during the 10 seconds.
Change in Function in Sitting Test for people with SCI (FIST-SCI) | baseline, up to 2 months
  FIST-SCI is a clinical test that will be used to test seated balance. FIST-SCI consists of 14 functional, everyday activities as test items. The items are scored on a 5 point ordinal scale ranging from 0 to 4, with 0 representing the lowest ability and 4 representing normal ability.
Change in Motor Evoked Potential (MEP) | baseline, up to 2 months
  MEP evaluates corticospinal excitability (strength of the connections between the brain and the muscles). The excitability is measured as a peak-to-peak amplitude in millivolts (mV).

CONTACTS AND LOCATIONS:
Overall Officials: Matija Milosevic, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No